CLINICAL TRIAL: NCT03508336
Title: The Initiation of Swallowing Can Indicate the Prognosis of Disorders of Consciousness
Brief Title: The Initiation of Swallowing Can Indicate the Prognosis of DOC
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Dr, Hangzhou Normal University
Other Study IDs: 2017A02529
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Minimally Conscious State; Vegetative State
Keywords: disorders of consciousness; swallowing; prognosis prediction; minimally conscious state; vegetative state
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with disorders of consciousness: Patients with disorders of consciousness from several brain injury, assessed by Coma Recovery Scale-Revised (CRS-R), have been clinically classified into coma, unresponsive wakefulness syndrome and minimally conscious state.
  Interventions: Diagnostic Test: Coma Recovery Scale-Revised

INTERVENTIONS:
Diagnostic Test: Coma Recovery Scale-Revised — Patients with disorders of consciousness were assessed by Coma Recovery Scale-Revised (CRS-R). In addition, we selected four stimuli: 1) only a command (as recommended in CRS-R), which was "open your mouth"; 2) only a spoon without a command; 3) a spoon and a command, the command was "there is a spoon and open your mouth"; 4) a spoon with water and a command, the command was "there is a spoon with water and open your mouth". In brief, we presented these stimuli orderly in front of the patient's mouth and presented any one of them over 4 trials at 15 second intervals.

SUMMARY:
This study is aimed to detect the initiation of swallowing act in DOC patients, to find if it is a good item as a stimulus and to detect the relationship between the initiation of swallowing act and the prognosis of DOC patients.

DETAILED DESCRIPTION:
Studies suggest that the initiation and patterning of swallowing of the pharyngeal phase is also under active cortical control for both spontaneous as well as volitional swallowing in awake humans and non-human primates. A recent study found that most patients of disorders of consciousness (DOC) would recover their swallowing ability quickly. And there is no study about detecting the initiation of swallowing act in DOC patients. This study is aimed to detect the initiation of swallowing act in DOC patients, to find if it is a good item as a stimulus and to detect the relationship between the initiation of swallowing act and the prognosis of DOC patients. DOC patients were recruited (standard diagnosis procedure is 4 times CRS-R testing within 2 weeks). The different four stimuli were as follows: 1) One command (as recommended in CRS-R) which was "open your mouth". 2) Put a spoon in front of the patient's mouth without a command. 3) One command with a spoon in front of the mouth, the command is "there is a spoon and open your mouth". 4) One command with a spoon full of water in front of the mouth, the command is "there is a spoon with water and open your mouth". We presented these stimuli orderly in front of the patient's mouth and presented any one of them over 4 trials at 15 second intervals.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* no administration of central nervous system stimulant, neuro-muscular blocking agents, or sedative within the prior 24 hours
* a diagnosis of VS or MCS-, based on the behavioral assessment of standardized CRS-R
* periods of eye opening (indicating preserved sleep-wake cycles).

Exclusion Criteria:

* documented history of prior brain injury
* premorbid illness resulting in documented functional disabilities up to time of the injury
* acute illness (e.g., pyrexia, pneumonia, diarrhea)
* receiving hyperbaric oxygen treatments within 2 hours
* fracture of the mandible.

Ages: 27 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with disorders of consciousness
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised （CRS-R） | Six month later
  examine the prognostic value of patients, longitudinal behavioral assessments were repeatedly conducted by means of the CRS-R 6-month later

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro, Study Chair — International Vegetative State and Consciousness Science Institute, Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Giacino JT, Schnakers C, Rodriguez-Moreno D, Kalmar K, Schiff N, Hirsch J. Behavioral assessment in patients with disorders of consciousness: gold standard or fool's gold? Prog Brain Res. 2009;177:33-48. doi: 10.1016/S0079-6123(09)17704-X. PMID 19818893
- [Background] Hansen TS, Engberg AW, Larsen K. Functional oral intake and time to reach unrestricted dieting for patients with traumatic brain injury. Arch Phys Med Rehabil. 2008 Aug;89(8):1556-62. doi: 10.1016/j.apmr.2007.11.063. PMID 18674990
- [Derived] Wang J, Wang J, Hu X, Xu L, Tian J, Li J, Fang D, Huang W, Sun Y, He M, Laureys S, Di H. The Initiation of Swallowing Can Indicate the Prognosis of Disorders of Consciousness: A Self-Controlled Study. Front Neurol. 2019 Nov 14;10:1184. doi: 10.3389/fneur.2019.01184. eCollection 2019. PMID 31798516